CLINICAL TRIAL: NCT03583502
Title: Maternal Supplementation With Krill Oil During Lactation: Effects on Human Milk Long-chain Polyunsaturated Fatty Acids
Brief Title: Krill Oil Supplementation: Effects on Breast Milk Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SO-2016-Krilling
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Breast Milk Expression
Keywords: LCPUFA; DHA; krill oil; supplementation; breast milk
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented (Experimental): krill oil and fish oil supplement
  Interventions: Dietary Supplement: krill oil and fish oil supplement
- Controls (No Intervention): The control group did not receive any supplementation.

INTERVENTIONS:
Dietary Supplement: krill oil and fish oil supplement — Administration of 2 gelatin soft capsules per day of a combined krill and fish oil supplement, providing 250 mg/day of DHA and 70 mg/day of EPA, for overall 30 days.
  Arms: Supplemented

SUMMARY:
Docosahexaenoic acid (DHA) belongs to long-chain polyunsaturated fatty acids (LCPUFAs) category and is a major building block for neuronal and retinal membranes, playing a crucial role in brain and visual development within the first months of life. Due to the lack of enzymes for the synthesis of its precursors, neonates strictly rely on dietary intakes of DHA. Antarctic krill (Euphausia superba) is a small crustacean rich in phospholipid-bound DHA, which is highly bioavailable, but whether it is effective in increasing DHA excretion in breast milk (BM) has not been investigated yet.

This study aims to evaluate whether maternal supplementation with krill oil during breastfeeding increases DHA contents in breast milk BM.

Mothers of infants admitted to the Neonatal Intensive Care Unit will be enrolled in this open, randomized, controlled study and randomly allocated in 2 groups. Group 1 will receive an oral krill oil-based supplement providing 250 mg/day of DHA and 70 mg/day of EPA for 30 days, whereas group 2 serves as control. BM samples from both groups will be collected at baseline (T0) and day 30 (T1) and will undergo a qualitative analysis of LCPUFAs composition by gas chromatography/mass spectrometry.

DETAILED DESCRIPTION:
Long-chain polyunsaturated fatty acids (LCPUFAs), such as docosahexaenoic (DHA, 22:6 n-3) and arachidonic acid (AA, 20:4 n-6), are major building blocks for the lipid bilayer of neuronal and retinal membranes. Brain maturation and visual development start during pregnancy and continue throughout the first year of life; hence, the role of LCPUFAs is greatest during this period.

Like all mammals, humans lack enzymes for the synthesis of n-3 and n-6 precursors of DHA and AA, which are therefore essential fatty acids and need to be provided by dietary sources.

Breast milk (BM) is the first nutritional choice in term and preterm neonates, and is considered an appropriate and natural source of essential fatty acids in this population. Among LCPUFAs, the role of DHA in the early phases of life has gained increased attention over the last 20 years. Several studies have proved the beneficial effects of DHA on visual acuity and learning skills in neonates; some of these trials have also underpinned the importance of dietary DHA sources, showing improved visual acuity in breastfed term neonates or preterm neonates fed LCPUFA-supplemented formula.

The amount of LCPUFAs excreted in BM, however, is significantly influenced by the related maternal dietary intakes, and this is particularly evident for mothers with extremely high fish consumption or on a vegetarian diet.

Sherry et al. have demonstrated that a 6-week supplementation with low or high dose of DHA in lactating women significantly increases DHA concentration in BM and maternal plasma compared with placebo; consistently, breastfed infants of supplemented mothers showed higher plasma DHA levels.

Antarctic krill, a small crustacean belonging to the order Euphausiacea, is by far the most dominant member of the Antarctic zooplankton community, and also represents a rich source of n-3 LCPUFAs, such as DHA and eicosapentaenoic acid (EPA). Compared to fish oil, krill oil has similar DHA contents, but provides higher amounts of EPA. In addition, fish oil fatty acids are mainly stored as triglycerides (TG), whereas in krill oil are predominantly incorporated to phospholipids (PL), with significantly enhanced bioavailability. To date, the effects of maternal supplementation with krill oil during lactation on BM LCPUFAs composition is still an issue for discussion/has not been investigated.

The aim of this pilot study is to evaluate whether oral maternal supplementation with krill oil combined to fish oil in breastfeeding mothers increases BM concentration of DHA.

Breastfeeding mothers of infants admitted to the Neonatal Intensive Care Unit of Sant'Orsola-Malpighi University Hospital, Bologna, Italy, will be consecutively enrolled if a written informed consent to participate in the present study is obtained.

Women enrolled will undergo open randomization to 2 groups. Group 1 will receive 2 gelatin soft capsules per day of a combined krill and fish oil supplement (Krilling D®, Italchimici S.P.A., Milan, Italy), providing 250 mg/day of DHA and 70 mg/day of EPA, for overall 30 days, whereas group 2 will serve as control. Ten ml of fresh mid-BM samples will be collected at baseline (T0) and at day 30 (T1) of supplementation in both groups.

After collection, DHA, AA and EPA contents of BM samples will be analyzed at the laboratory of the Center for Applied Biomedical Research (CRBA) of Sant'Orsola-Malpighi University Hospital, Bologna, Italy, using gas chromatography/mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

- ongoing breastfeeding

Exclusion Criteria:

- ongoing LCPUFA supplementation at the time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Breast milk excretion of docosahexaenoic acid (DHA) | Baseline (T0)
  Qualitative analysis of DHA concentration in breast milk
Breast milk excretion of docosahexaenoic acid (DHA) | After 30 days of supplementation (T1)
  Qualitative analysis of DHA concentration in breast milk

SECONDARY OUTCOMES:
Breast milk excretion of eicosapentaenoic acid (EPA) | Baseline (T0)
  Qualitative analysis of EPA concentration in breast milk
Breast milk excretion of eicosapentaenoic acid (EPA) | After 30 days of supplementation (T1)
  Qualitative analysis of EPA concentration in breast milk
Breast milk excretion of arachidonic acid (AA) | Baseline (T0)
  Qualitative analysis of AA concentration in breast milk
Breast milk excretion of arachidonic acid (AA) | After 30 days of supplementation (T1)
  Qualitative analysis of AA concentration in breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Corvaglia, Prof, Principal Investigator — luigi.corvaglia@unibo.it
Locations (1):
- Neonatal Intensive Care Unit of the S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cimatti AG, Martini S, Munarini A, Zioutas M, Vitali F, Aceti A, Mantovani V, Faldella G, Corvaglia L. Maternal Supplementation With Krill Oil During Breastfeeding and Long-Chain Polyunsaturated Fatty Acids (LCPUFAs) Composition of Human Milk: A Feasibility Study. Front Pediatr. 2018 Dec 20;6:407. doi: 10.3389/fped.2018.00407. eCollection 2018. PMID 30622936